CLINICAL TRIAL: NCT00792051
Title: A Randomised Controlled Trial of the Effectiveness of Vaccinating Children to Reduce Household Transmission of Influenza
Brief Title: Direct and Indirect Benefits of Influenza Vaccine Versus Placebo in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Fund for the Control of Infectious Diseases (Unknown); Research Grants Council, Hong Kong (Other); Centre for Health Protection, Hong Kong (Other Government)
Responsible Party: Dr Benjamin John Cowling, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GML003.4
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Influenza Virus Infection
Keywords: influenza; vaccination; children; Influenza-like illness
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Influenza vaccine
  Interventions: Biological: Inactivated influenza vaccine
- 2 (Placebo Comparator)
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Inactivated influenza vaccine — 0.5ml intramuscular single dose
  Other Names: VAXIGRIP®, Sanofi Pasteur
  Arms: 1
Biological: Saline — 0.5ml intramuscular, one dose
  Arms: 2

SUMMARY:
While immunisation of school-age children against influenza is not recommended in Hong Kong, past experience in Japan and elsewhere suggests that immunisation of children may protect the wider community through its indirect transmission-limiting impact as well as the direct immunologic protection afforded vaccinated children themselves. We aim to assess whether vaccinating children against influenza protects vaccinees as well as their household contacts from infection.

DETAILED DESCRIPTION:
Design and subjects: A double-blind randomised controlled trial of 800 subjects aged 6-17 drawn from the general population and their 2000 household contacts. The subjects will be randomised in a 3:2 ratio to the intervention and placebo groups, respectively. Serum samples will be collected from subjects pre- and 1 month post-vaccination, and after the influenza season. Serum samples will be collected from household contacts at baseline and at the end of the influenza season. During the follow-up period, subjects and household members will keep symptom diaries and those reporting influenza-like-illness will be offered free doctor consultations or home visits where we will arrange for collection of nose and throat swabs.

Study instruments: An antibody titre of ≥40 in the post-vaccine serum will be used to define seroprotection to those particular strains, while a four-fold or higher increase in antibody titres between baseline and end-of-season follow-up of the household contacts will define influenza infection during the season. Subjects and household contacts will be asked to keep symptom diaries, and during episodes of ILI we will collect nose and throat swabs for laboratory confirmation of influenza infection; the primary serology results will then be compared with clinical and laboratory-confirmed influenza episodes.

Interventions: 1 (intervention) inactivated influenza vaccine (Vaxigrip, Sanofi Pasteur); 2 (placebo) saline injection.

Main outcome measures: The proportions of subjects and household contacts with serology-confirmed influenza infection during follow-up among the 2 intervention arms.

Analysis: Intention to treat, adjusting for within-household correlation in influenza attack rates.

ELIGIBILITY:
Inclusion Criteria:

* All vaccinees must be Hong Kong residents aged between 6 and 17.

Exclusion Criteria:

* Vaccinees should not be allergic or hypersensitive to the active substances or components (eggs, chicken proteins, formaldehyde, neomycin, etc.) used in the vaccines or where vaccination is otherwise contraindicated. Subjects should not have an underlying immunocompromised condition or be receiving immunosuppressive agents.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The proportions of subjects and household contacts with serology-confirmed influenza infection during follow-up among the 2 intervention arms. | nine months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Cowling, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Result] Cowling BJ, Ng S, Ma ES, Fang VJ, So HC, Wai W, Cheng CK, Wong JY, Chan KH, Ip DK, Chiu SS, Peiris JS, Leung GM. Protective efficacy against pandemic influenza of seasonal influenza vaccination in children in Hong Kong: a randomized controlled trial. Clin Infect Dis. 2012 Sep;55(5):695-702. doi: 10.1093/cid/cis518. Epub 2012 Jun 5. PMID 22670050
- [Result] Cowling BJ, Ng S, Ma ES, Cheng CK, Wai W, Fang VJ, Chan KH, Ip DK, Chiu SS, Peiris JS, Leung GM. Protective efficacy of seasonal influenza vaccination against seasonal and pandemic influenza virus infection during 2009 in Hong Kong. Clin Infect Dis. 2010 Dec 15;51(12):1370-9. doi: 10.1086/657311. Epub 2010 Nov 10. PMID 21067351
- [Derived] Cowling BJ, Perera RA, Fang VJ, Chan KH, Wai W, So HC, Chu DK, Wong JY, Shiu EY, Ng S, Ip DK, Peiris JS, Leung GM. Incidence of influenza virus infections in children in Hong Kong in a 3-year randomized placebo-controlled vaccine study, 2009-2012. Clin Infect Dis. 2014 Aug 15;59(4):517-24. doi: 10.1093/cid/ciu356. Epub 2014 May 13. PMID 24825868